CLINICAL TRIAL: NCT04295577
Title: Multi-Centre Observational Study of Maintenance Niraparib in Treatment of Ovarian CanceR: UK Routine Clinical Practice Experience
Brief Title: Multi-Centre Observational Study of Maintenance Niraparib in Treatment of Ovarian CanceR
Acronym: MONITOR-UK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR4939
Record Dates: First submitted 2020-01-13; First posted 2020-03-04 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer
Keywords: Niraparib
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — niraparib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Cohort 1: Retrospective Cohort: This cohort will include:
  * Patients who have previously commenced maintenance Niraparib prior to the MONITOR study opening at the site and are still receiving Niraparib but in whom quality of life data are not available.
  * Patients who have previously commenced Niraparib prior to the MONITOR Study opening at the site but are now deceased but will be eligible for retrospective data collection without the need for informed consent.
  * Patients who have previously commenced maintenance Niraparib prior to the MONITOR study opening at the site but have discontinued treatment.
  * Data in respect of AEs, SAEs, ADRs and AESIs will be recorded in Case Report Forms and be identified via the patient's medical records. There is no requirement to complete trial specific SAE reporting forms in this cohort.
  Interventions: Other: Niraparib
- Cohort 2: Prospective Cohort: This cohort will include:
  * Patients who have previously commenced maintenance Niraparib prior to the MONITOR study opening at the site and are still receiving Niraparib and in whom quality of life data is available.
  * Patients who are due to commence maintenance Niraparib treatment.
  Interventions: Other: Niraparib

INTERVENTIONS:
Other: Niraparib — Niraparib - Niraparib is an oral, highly selective PARP-1 and -2 inhibitor. However, it also inhibits other members of the PARP family, including PARP 3, -4, -10, 12, -14, and -15[13].

SUMMARY:
This is a multi-centre, observational (non-interventional) study, designed to follow patients with advanced ovarian fallopian tube and primary peritoneal cancer, who are receiving Niraparib as maintenance treatment, according to the Niraparib access criteria (via TESARO patient access programme, EMA licence and NHS pending NICE assessment due 2018) including assessment of tolerability to Niraparib therapy.

DETAILED DESCRIPTION:
This is a multi-centre, observational (non-interventional) study, designed to follow patients with advanced ovarian fallopian tube and primary peritoneal cancer, who are receiving Niraparib as maintenance treatment, according to the Niraparib access criteria (via TESARO patient access programme, EMA licence and NHS pending NICE assessment due 2018) including assessment of tolerability to Niraparib therapy. These pathways will include patients who have been registered and not prescribed drug. In these cases, the reason for patients not receiving Niraparib will be recorded. Up to 16 centres will be involved in the study. Centres will be selected based on interest in or experience of prescribing Niraparib and geographical location in order to give a representative picture of the management of Niraparib in the UK.

Cohort 1: Retrospective Cohort

This cohort will include:

* Patients who have previously commenced maintenance Niraparib prior to the MONITOR study opening at the site and are still receiving Niraparib but in whom quality of life data are not available.
* Patients who have previously commenced Niraparib prior to the MONITOR Study opening at the site but are now deceased but will be eligible for retrospective data collection without the need for informed consent.
* Patients who have previously commenced maintenance Niraparib prior to the MONITOR study opening at the site but have discontinued treatment.
* Data in respect of AEs, SAEs, ADRs and AESIs will be recorded in Case Report Forms and be identified via the patient's medical records. There is no requirement to complete trial specific SAE reporting forms in this cohort.

Cohort 2: Prospective Cohort

This cohort will include:

* Patients who have previously commenced maintenance Niraparib prior to the MONITOR study opening at the site and are still receiving Niraparib and in whom quality of life data is available.
* Patients who are due to commence maintenance Niraparib treatment.

The collection of QoL data, using EQ-5D-5L and EORTC QoL-OV28, FACT-O questionnaires will be mandatory. For patients continuing on Niraparib, data will be collected retrospectively to the point they sign the consent form, and prospectively. Going forward QoL data will not be collected for these patients unless available as part of routine clinical care and baseline QoL is available.

The collection of data relating to adverse events will be mandatory. The scope of adverse events to be recorded includes AEs, SAEs, ADRs and AESIs - see section 5.3.1 for definitions of these events. Details in respect of AEs and SAEs, ADRs and AESIs will be recorded during routine clinic visits or via standard of care contact with the patient.

No additional visits will be required, no study medication will be administrated, and no additional procedures will be performed outside the local routine practice as part of the trial. Patients will be managed and followed up according to routine practice. Only data available in the patient's medical record will be collected. Patients consented to cohort 2 will be asked to complete validated QoL tools; EQ-5D-5L, FACT-O and EORTC QOL-OV28. Approximately 350 patients will be enrolled with an estimated 100 in the retrospective cohort and 250 in the prospective cohort.

ELIGIBILITY:
Inclusion Criteria:

* Female patient 18 years old or over
* Patients who are planned to receive Niraparib for advanced ovarian fallopian tube or primary peritoneal cancer,
* Patients who have previously commenced maintenance Niraparib prior to study opening at site
* Deceased patients who have previously been prescribed Niraparib
* Patients able to give written informed consent, complete questionnaires in English and comply with study procedures (if applicable).

Exclusion Criteria:

* Patients aged <18 years old
* Patients unable to give informed consent, complete questionnaires in English or comply with study procedures (if applicable).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: Patients with advanced ovarian fallopian tube and primary peritoneal cancer, who are/have/ will be receiving Niraparib as maintenance treatment
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2024-02-03 (Estimated); Study Completion 2024-02-03 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events | February 2020 - August 2022
  Proportion of patients with at least one grade ≥3 treatment emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Treatment history for patients on Niraparib maintenance treatment | February 2020 - February 2024
  This will be composed of previous treatment details including duration, delays/ dose modifications.
Patient demographics for patients on Niraparib maintenance treatment | February 2020 - February 2024
  To describe the patient population of those on Niraparib.
Medical history for patients on Niraparib maintenance treatment | February 2020 - February 2024
  To ascertain the rationale for patients receiving Niraparib maintenance therapy
Routine clinical practice of Niraparib maintenance treatment | February 2020 - February 2024
  To detail clinical management of Niraparib maintenance therapy in a real-world pragmatic setting.
Time to First Subsequent Therapy (TFST) | February 2020 - February 2024
  This will be defined as the date of the start of Niraparib to the start date of the first subsequent anticancer therapy. The treatment prescribed at TFST will also be recorded.
Chemotherapy Free Interval (CFI) | February 2020 - February 2024
  This will be defined as the time from the last platinum-based chemotherapy dose until initiation of next anticancer therapy (excluding maintenance therapy).
Objective Response Rate (ORR) | February 2020 - February 2024
  Where indicated for Niraparib treatment, only for patients with measurable disease on baseline imaging. This will be defined as complete or partial response as judged by the investigator.
Progression Free Survival (PFS) | January 2022 - February 2024
  This will be defined as time from start of Niraparib treatment to progression or death from any cause. Patients without an event will be censored at day of last follow up. Progression will be assessed by the investigator according to routine practice
Quality of life for patients on Niraparib maintenance treatment | February 2020 - February 2024
  Quality of life (QoL) at protocol-specified time points will be assessed.
Adverse events for patients on Niraparib maintenance treatment | February 2020 - February 2024
  Number of Adverse Events (AEs), Adverse Drug Reactions (ADRs), Serious Adverse Events (SAEs) and Averse Events of Special lnterest (AESIs)

CONTACTS AND LOCATIONS:
Overall Officials: Susana Banerjee, MBBS MA PhD FRCP, Study Chair — Royal Marsden NHS Foundation Trust
Locations (15):
- United Kingdom (15):
  - Royal United Hospitals Bath, Bath
  - Belfast Health & Social Care Trust, Belfast
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - University Hospitals Bristol NHS Foundation Trust, Bristol
  - Addenbrookes Hospital, Cambridge
  - Velindre Cancer Centre, Velindre University NHS Trust, Cardiff
  - Morecambe Bay NHS Trust, Lancaster
  - St James's University Hospital, Leeds
  - Barts Health NHS Trust, London
  - Northampton General Hospital NHS Trust, Northampton
  - Mount Vernon Cancer Centre, East and North Hertfordshire NHS Trust, Northwood
  - Queen's Hospital, Romford
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Royal Marsden NHS Foundation Trust, Sutton
  - Royal Cornwall Hospitals NHS Trust, Truro

IPD SHARING:
Plan to Share IPD: No